CLINICAL TRIAL: NCT01492920
Title: A Randomized, Double-Blinded, Placebo Controlled Phase III Trial Using Acetyl-L-Carnitine(ALC)(NSC# 747431) for the Prevention of Chemotherapy-Induced Peripheral Neuropathy in Patients With Recurrent Ovarian, Primary Peritoneal or Fallopian Tube Cancer
Brief Title: Acetyl-L-Carnitine Hydrochloride in Preventing Peripheral Neuropathy in Patients With Recurrent Ovarian Epithelial Cancer, Primary Peritoneal Cavity Cancer, or Fallopian Tube Cancer Undergoing Chemotherapy
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Withdrawn
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: GOG-0257; NCI-2012-00090 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000719317; GOG-0257 (Other: Gynecologic Oncology Group); GOG-0257 (Other: DCP); GOG-0257 (Other: CTEP); U10CA101165 (NIH)
Record Dates: First submitted 2011-12-14; First posted 2011-12-15 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Fatigue; Malignant Ovarian Mixed Epithelial Tumor; Neuropathy; Neurotoxicity Syndrome; Ovarian Brenner Tumor; Ovarian Clear Cell Cystadenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Mucinous Cystadenocarcinoma; Ovarian Serous Cystadenocarcinoma; Pain; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fatigue; Neurotoxicity Syndromes; Brenner Tumor; Pain; Fallopian Tube Neoplasms; Ovarian Neoplasms

ARMS (2):
- Arm I (acetyl-L-carnitine hydrochloride) (Experimental): Patients receive ALC PO BID on days 1-21 (during chemotherapy treatment).
  Interventions: Dietary Supplement: Acetyl-L-Carnitine Hydrochloride; Other: Questionnaire Administration; Other: Quality-of-Life Assessment
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO BID on days 1-21 (during chemotherapy treatment) (maximum of 8 courses).
  Interventions: Other: Placebo; Other: Questionnaire Administration; Other: Quality-of-Life Assessment

INTERVENTIONS:
Dietary Supplement: Acetyl-L-Carnitine Hydrochloride — Given orally
  Other Names: Acetylcarnitine Hydrochloride, L-; Acetylcarnitine L-form HCl
  Arms: Arm I (acetyl-L-carnitine hydrochloride)
Other: Placebo — Given orally
  Other Names: PLCB
  Arms: Arm II (placebo)
Other: Questionnaire Administration — Ancillary studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This randomized phase III trial studies how well acetyl-L-carnitine hydrochloride works compared to a placebo in preventing peripheral neuropathy in patients with recurrent ovarian epithelial cancer, primary peritoneal cancer, or fallopian tube cancer undergoing chemotherapy. Acetyl-L-carnitine hydrochloride may prevent or lessen peripheral neuropathy caused by chemotherapy. It is not yet known whether acetyl-L-carnitine hydrochloride is more effective compared to a placebo in preventing peripheral neuropathy caused by chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the therapeutic efficacy of acetyl-L-carnitine hydrochloride (ALC) in preventing chemotherapy-induced peripheral neuropathy (CIPN) in patients with recurrent ovarian, primary peritoneal, or fallopian tube cancer.

SECONDARY OBJECTIVES:

I. Evaluate the effect of ALC on chemotherapy-induced fatigue based upon the Functional Assessment of Cancer Therapy (FACT)-Fatigue scale.

II. Evaluate the effect of ALC on sensory peripheral neuropathy as measured with the first 4 items of the FACT/Gynecologic Oncology Group (GOG)-Neurotoxicity (Ntx) subscale (FACT/GOG-Ntx_4 subscale).

III. Evaluate the effect of ALC on the health-related quality of life as measured by the FACT-Ovarian (O) trial outcome index (TOI).

OUTLINE: This is a multicenter study. Patients are stratified according to planned dosage of paclitaxel (< 150 mg/m^2 vs ≥ 150 mg/m^2), and age (< 60 years of age vs ≥ 6 years of age). Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive acetyl-L-carnitine hydrochloride (ALC) orally (PO) twice daily (BID) on days 1-21 (during chemotherapy treatment).

ARM II: Patients receive placebo PO BID on days 1-21 (during chemotherapy treatment) (maximum of 8 courses).

In both arms, treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

Patients also complete questionnaires comprising the Functional Assessment of Cancer Therapy (FACT)-Fatigue scale, the FACT-Gynecologic Oncology Group Neurotoxicity subscale (FACT/GOG-Ntx_4 subscale), and the FACT-Ovarian trial outcome index (FACT-O TOI) at baseline, prior to courses 3 and 5, within 4 weeks after completion of treatment, and then at 3 months after completion of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologic diagnosis of epithelial ovarian carcinoma, peritoneal primary or fallopian tube carcinoma, which is now recurrent
* Patients with the following histologic epithelial cell types are eligible: serous adenocarcinoma, endometrioid adenocarcinoma, mucinous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, transitional cell carcinoma, malignant Brenner tumor, or adenocarcinoma not otherwise specified (N.O.S.)
* All patients must have had a treatment-free interval without clinical evidence of progressive disease of at least 6 months from completion of front-line chemotherapy (both platinum and taxane); front-line therapy may have included a biologic agent (i.e., bevacizumab)

  * Front-line treatment may include maintenance therapy following complete clinical or pathological response; however, maintenance cytotoxic chemotherapy must be discontinued for a minimum of 6 months prior to documentation of recurrent disease; patients receiving maintenance biological therapy or hormonal therapy are ELIGIBLE provided their recurrence is documented more than 6 months from primary cytotoxic chemotherapy completion (includes maintenance chemotherapy) AND a minimum 4 weeks has elapsed since their last infusion of biological therapy
  * Patients receiving hormonal therapy for biochemical or non-measurable recurrence disease are ELIGIBLE provided their recurrence is documented more than 6 months following the completion of primary cytotoxic chemotherapy; a minimum of 4 weeks must have expired since their last exposure to hormonal therapy

    * The complete response to front-line chemotherapy must have included a negative physical exam, normalization of CA125 if elevated at baseline, and negative radiographic assessment of disease, if obtained
    * Patients who have undergone reassessment laparotomy or laparoscopy following primary therapy are eligible for this study as long as they demonstrated a pathologic complete response based on the surgical assessment (i.e. all obtained specimens were histologically negative for disease)
* Patients with a past history of primary endometrial cancer within the last five years are excluded unless all of the following conditions are met:

  * Stage not greater than IB
  * No more than superficial myometrial invasion, without vascular or lymphatic invasion
  * No poorly differentiated subtypes, including papillary serous, clear cell, or other International Federation of Gynecology and Obstetrics (FIGO) grade 3 lesions
* Patients must be expected to receive a minimum of 2 cycles of paclitaxel and a platinating agent for their recurrent disease;

  * Addition of other drugs such as bevacizumab is acceptable as long as these additional drugs are not typically associated with peripheral neuropathy
  * The initial, planned infusion duration of each dose of paclitaxel must be 3 hours or less
* Patients must start the study with a GOG performance status of 2 or less
* Serum creatinine ≤ 2.5 mg/dL
* Neuropathy (sensory and motor) less than or equal to the National Cancer Institute (NCI) CTCAE v4.0 grade 1
* No patients with a history of seizure activity
* No patients who are unable to swallow oral medications
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer, are excluded if there is any evidence of other malignancy being present within the last five years
* No patients of childbearing potential not practicing adequate contraception
* No patients who are pregnant or nursing
* No patients who are known to have diabetes
* No patients with known allergies to ALC (acetyl-L-carnitine hydrochloride)
* Patients are excluded if their previous cancer treatment contraindicates this protocol therapy
* No patients who have received more than one previous regimen of chemotherapy (maintenance is not considered a second regimen)
* No patients receiving concurrent immunotherapy or radiotherapy
* No patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis
* No patients who are currently receiving or have received warfarin or acenocoumarol within the past 7 days
* No patients taking > 100 units of racemic vitamin E (or > 50 units of ααα-tocopherol) daily within 5 days of starting study therapy
* No patients taking other medications (Rx, OTC, or dietary supplements) to prevent or treat neuropathy within 5 days of starting study treatment; such products include:

  * Gabapentin (Neurontin ®)
  * Pregabalin (Lyrica ®)
  * Duloxetine (Cymbalta ®)
  * Alpha-lipoic acid
  * Note that tricyclic antidepressants or selective serotonin/norepinephrine-selective reuptake inhibitors prescribed for the treatment of mood disorders are allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Chemotherapy-related peripheral neuropathy as measured with Functional Assessment of Cancer Therapy (FACT)/GOG-Ntx subscale | Up to 3 months

SECONDARY OUTCOMES:
Chemotherapy-related fatigue as measured with FACT-Fatigue | Up to 3 months
Patient-reported sensory peripheral neuropathy, as measured by the FACT/GOG-Ntx v4 subscale | Up to 3 months
Quality of life, as measured by the FACT-O TOI | Up to 3 months
  Tested at significance level of 5%.

CONTACTS AND LOCATIONS:
Overall Officials: David Kushner, Principal Investigator — Gynecologic Oncology Group